CLINICAL TRIAL: NCT06592924
Title: A Randomized Phase III Clinical Trial for the Addition of Docetaxel to Androgen Receptor Pathway Inhibitors in Patients With Metastatic Castration Sensitive Prostate Cancer and Suboptimal PSA Response
Brief Title: Docetaxel to Androgen Receptor Pathway Inhibitors in Patients With Metastatic Castration Sensitive Prostate Cancer and Suboptimal PSA Response
Acronym: TRIPLE-SWITCH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: ECOG-ACRIN Cancer Research Group (Network); NRG Oncology (Other); Alliance for Clinical Trials in Oncology (Other); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCTG-PR26; CCTG-PR26 (Other: NCI/CTEP); NCI-2024-07535 (Other: NCI CTRP)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: PR26; Castration sensitive
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — abiraterone; enzalutamide; apalutamide; darolutamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard ADT + ARPI (Active Comparator)
  Interventions: Drug: Abiraterone; Drug: Enzalutamide; Drug: Apalutamide; Drug: Darolutamide (BAY 1841788); Drug: ADT
- Docetaxel + Standard ADT + ARPI (Experimental)
  Interventions: Drug: Abiraterone; Drug: Enzalutamide; Drug: Apalutamide; Drug: Darolutamide (BAY 1841788); Drug: Docetaxel; Drug: ADT

INTERVENTIONS:
Drug: Abiraterone — Assigned prior to enrollment
Drug: Enzalutamide — Assigned prior to enrollment
Drug: Apalutamide — Assigned prior to enrollment
Drug: Darolutamide (BAY 1841788) — Assigned prior to enrollment
Drug: Docetaxel — Assigned at enrollment
  Arms: Docetaxel + Standard ADT + ARPI
Drug: ADT — Physician's choice. Assigned prior to enrollment

SUMMARY:
This study is being done to answer the following question: can the chance of prostate cancer growing or spreading be lowered by adding a drug to the usual combination of drugs?

This study would like to find out if this approach is better or worse than the usual approach for prostate cancer.

The usual approach for patients who are not in a study is hormone treatment with Androgen Deprivation Therapy (ADT) and Androgen-Receptor Pathway Inhibitor (ARPI).

DETAILED DESCRIPTION:
This is an international multi-centre, open-label, randomized phase III trial comparing Docetaxel chemotherapy added to standard of care Androgen Deprivation Therapy (ADT) + Androgen-Receptor Pathway Inhibitor (ARPI) versus standard of care Androgen Deprivation Therapy (ADT) + Androgen-Receptor Pathway Inhibitor (ARPI) in participants with metastatic castration sensitive prostate cancer (mCSPC) who have a suboptimal PSA response after 6-12 months of androgen-targeting therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed adenocarcinoma of the prostate
* Metastatic disease by conventional imaging
* PSA of ≥5.0 ng/ml (5.0 ug/L) prior to commencement of ADT
* Receipt of ADT for mCSPC for at least 6 months and no greater than 12 months at time of enrollment.
* Receipt of ARPI (e.g. abiraterone acetate, enzalutamide, apalutamide, or darolutamide) for at least 4 months at time of enrollment
* Potential trial participants should have recovered from clinically significant adverse events of their most recent therapy/intervention prior to enrollment.
* Serum testosterone <1.7 nmol/L or 50 ng/dL.
* PSA ≥ 0.2 ng/ml (0.2 ug/L) within 14 days of enrollment. If there is any rise in PSA since starting ADT and achieving castrate-level testosterone, PSA must be repeated and must not fulfill ineligibility criteria 4.2.1.
* Candidate for docetaxel chemotherapy
* ECOG Performance Status (PS) 0 to 2.
* Adequate organ and marrow function measured within 14 days prior to enrollment.
* Participant consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each participant must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Participants must be accessible for treatment and follow-up. Investigators must assure themselves the participants enrolled on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* In accordance with CCTG policy, protocol treatment is to begin within 5 working days of participant enrollment.
* If the participant and the participant's partner are of childbearing potential, they must agree to use medically accepted methods of contraception
* HIV-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Participant access to all protocol therapies must be confirmed prior to enrollment

Exclusion Criteria:

* Two consecutive rises in PSA since achieving castration on ADT at least 2 weeks apart with at least one PSA ≥5% above the PSA nadir and with at least one PSA having an absolute increase of ≥0.5 ng/ml above the PSA nadir.
* Evidence of radiographic progression or clinical progression since start of ADT.
* Docetaxel criteria:

  * Prior treatment with taxane chemotherapy
  * Grade 2 or worse peripheral neuropathy
  * Severe hypersensitivity to drugs formulated with polysorbate 80
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better.
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make this protocol unreasonably hazardous.
* Patients with a prior or concurrent malignancy whose natural history of treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Concurrent treatment with other anti-cancer systemic therapy other than ADT and ARPI.
* Live attenuated vaccination administered within 30 days prior to enrollment/randomization.
* For participants with a history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* High-grade neuroendocrine prostate cancer or small cell features.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 830 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2031-03-14 (Estimated); Study Completion 2031-04-15 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 39 months

SECONDARY OUTCOMES:
PSA Progression compared in both arms | 39 months
PSA Response comparison between arms | 39 months
  PCWG3 criteria
PSA Kinetics compared between both arms | 39 months
  * 90% PSA decline
  * PSA <0.2ng/ml
  * PSA <0.02ng/ml
Clinical progression-free survival between both arms | 39 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ong, Study Chair — Ottawa Hospital Research Institute, Ottawa ON Canada; Alexandra Sokolova, Study Chair — Oregon Health and Science University, Portland, OR, USA
Locations (310):
- United States (294):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Mercy Cancer Center, Merced, California
  - Providence Queen of The Valley, Napa, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Saint Joseph's Medical Center, Stockton, California
  - City of Hope South Bay, Torrance, California
  - City of Hope Upland, Upland, California
  - Woodland Memorial Hospital, Woodland, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - UCHealth - Cherry Creek, Denver, Colorado
  - Dillon Health Center/Shaw Cancer Center, Dillon, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - UCHealth Lone Tree Health Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Saint Anthony North Hospital, Westminster, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Springs, Coral Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - University of Miami Sylvester Comprehensive Cancer Center at Sole Mia, North Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Straub Medical Center - Kahului Clinic, Kahului, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Straub Pearlridge Clinic, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - University of Illinois, Chicago, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Pella, Pella, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Metairie, Metairie, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Veteran's Administration Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Allegiance Health, Jackson, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health - Baxter Clinic, Baxter, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Saint Joseph's Crosslake Clinic, Crosslake, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Essentia Health - Ely Clinic, Ely, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Essentia Health - Moose Lake Clinic, Moose Lake, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Essentia Health - Saint Joseph's Pequot Lakes Clinic, Pequot Lakes, Minnesota
  - Essentia Health - Saint Joseph's Pine River Clinic, Pine River, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health - Saint Joseph's Staples Clinic, Staples, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Hi-Line Sletten Cancer Center, Havre, Montana
  - Benefis Helena Specialty Center, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Hood River Memorial Hospital, Hood River, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Cancer Center Dickson City, Dickson City, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Philadelphia Veterans Administration Medical Center, Philadelphia, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Houston Methodist San Jacinto Hospital, Baytown, Texas
  - Houston Methodist Cypress Hospital, Cypress, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Richmond Community Hospital, Richmond, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - Tamarack Health Hayward Medical Center, Hayward, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Memorial Hospital of Laramie County, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
- Canada (16):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Waterloo Regional Health Network, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Niagara Health System-Saint Catharines General, Saint Catharines, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CSSS Champlain-Charles Le Moyne, Greenfield Park, Quebec
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHA Hopital L'Enfant-Jesus, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Access Criteria: Based on CCTG Policies
URL: https://www.ctg.queensu.ca/docs/public/policies/DataSharingandAccessPolicy.pdf